CLINICAL TRIAL: NCT04385667
Title: The Efficacy of Levonorgestrel Intrauterine System Versus Oral Megesterol Acetate in Treatment of Atypical Endometrial Hyperplasia. A Randomized Controlled Trial.
Brief Title: LVN- IUS Versus Oral Megesterol Acetate in Treatment of Atypical Endometrial Hyperplasia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hytham Atia, Associate Professor Obstetrics & Gynecology, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LVN-IUS vs Megace for AEH
Record Dates: First submitted 2020-05-09; First posted 2020-05-13 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Atypical Endometrial Hyperplasia
Keywords: atypical endometrial hyperplasia; levonorgestrel intrauterine system; Megestrol acetate; partial regression
MeSH Terms: conditions — Endometrial Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- levonorgestrel intrauterine system (LNG-IUD) (Active Comparator): levonorgestrel intrauterine system (LNG-IUD) applied.
  * Follow up endometrial sampling will be scheduled for all study patients in 3 months manner for at least one year. Specimens will be reviewed by single expert pathologist.
  * Patients with persistent atypical hyperplasia in specimens done after 6 months of start of therapy will be considered resistant to therapy and hysterectomy will be done.
  * Primary and secondary outcome data will be collected in tables with the other demographic data. All will be processed in tables for statistical analysis.
  Interventions: Device: levonorgestrel intrauterine system (LNG-IUD)
- Megestrol acetate (MA) (Active Comparator): Megesterol arm will receive 160 mg daily
  * Follow up endometrial sampling will be scheduled for all study patients in 3 months manner for at least one year. Specimens will be reviewed by single expert pathologist.
  * Patients with persistent atypical hyperplasia in specimens done after 6 months of start of therapy will be considered resistant to therapy and hysterectomy will be done.
  * Primary and secondary outcome data will be collected in tables with the other demographic data. All will be processed in tables for statistical analysis.
  Interventions: Drug: Oral Megesterol 160 mg daily

INTERVENTIONS:
Device: levonorgestrel intrauterine system (LNG-IUD) — progestin delivery for regression of atypical endometrial hyperplasia
  Other Names: • Follow up endometrial sampling will be scheduled for all study patients in 3 months manner for at least one year. Specimens will be reviewed by single expert pathologist.
  Arms: levonorgestrel intrauterine system (LNG-IUD)
Drug: Oral Megesterol 160 mg daily — progestin delivery for regression of atypical endometrial hyperplasia
  Other Names: • Follow up endometrial sampling will be scheduled for all study patients in 3 months manner for at least one year. Specimens will be reviewed by single expert pathologist.
  Arms: Megestrol acetate (MA)

SUMMARY:
This randomized controlled trial is aimed to compare the efficacy between Megestrol acetate (MA) and the levonorgestrel intrauterine system (LNG-IUD) regarding the ability and duration to produce complete regression for cases with atypical endometrial hyperplasia.

DETAILED DESCRIPTION:
Up to 25% of cases with endometrial cancer and atypical hyperplasia occur in premenopausal women. The progressively increasing trend of delay in first conception increases such patients who wish to have children.3 The recommended treatment for EH without atypia is primarily hormonal, whereas the preferred treatment for EH with atypia is hysterectomy given the significant risk for both concurrent and subsequent development of endometrial carcinoma. A dilemma results when EH with atypia is diagnosed in women who wish to retain fertility or declining doing hysterectomy due to concomitant medical morbidities. In these women, a trial of hormone therapy can be considered.4,5 In recent years, progestin therapy has been successfully used to treat selected women with endometrial cancer and atypical hyperplasia who desire to preserve fertility or having severe medical co-morbidities precluding (immediate) surgery. The most common progestin regimens include Megestrol acetate (MA) and the levonorgestrel intrauterine system (LNG-IUD).5-7

ELIGIBILITY:
Inclusion Criteria:

All cases with evidence of atypical endometrial hyperplasia declining doing hysterectomy

Exclusion Criteria:

* Cases with evidence of associated endometrial cancer.
* Cases with simple hyperplasia without atypia.
* Patients failed to collect at least 2 endometrial samples during treatment course.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-25 (Actual)

PRIMARY OUTCOMES:
The success rate to accomplish complete regression of atypical endometrial hyperplasia | 15 month
  The success rate to accomplish complete regression of atypical endometrial hyperplasia

SECONDARY OUTCOMES:
a- Duration needed to accomplish the complete recovery | 15 months
  time till regression
b- The partial regression and failure rates. | 8 months
  incidence of partial regression and therapy failure
c- Differential response rates between premenopausal and postmenopausal cases. | 15 months
  response rate in both premenopause and postmenopause women
d- The risk of thromboembolic complications | 15 months
  incidence of thromboembolism with therapy
f- Metabolic complications rates | 15 months
  occurence of diabetes or hypertension ...ets

CONTACTS AND LOCATIONS:
Overall Officials: Amr Alnemr, M.D., Principal Investigator — Faculty of Medicine- Zagazig university; Hytham Atia, M.D., Principal Investigator — Faculty of Medicine- Zagazig university
Locations (1):
- Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armstrong AJ, Hurd WW, Elguero S, Barker NM, Zanotti KM. Diagnosis and management of endometrial hyperplasia. J Minim Invasive Gynecol. 2012 Sep-Oct;19(5):562-71. doi: 10.1016/j.jmig.2012.05.009. Epub 2012 Aug 3. PMID 22863972
- [Background] Salman MC, Usubutun A, Boynukalin K, Yuce K. Comparison of WHO and endometrial intraepithelial neoplasia classifications in predicting the presence of coexistent malignancy in endometrial hyperplasia. J Gynecol Oncol. 2010 Jun;21(2):97-101. doi: 10.3802/jgo.2010.21.2.97. Epub 2010 Jun 30. PMID 20613899
- [Background] Zhou R, Yang Y, Lu Q, Wang J, Miao Y, Wang S, Wang Z, Zhao C, Wei L. Prognostic factors of oncological and reproductive outcomes in fertility-sparing treatment of complex atypical hyperplasia and low-grade endometrial cancer using oral progestin in Chinese patients. Gynecol Oncol. 2015 Dec;139(3):424-8. doi: 10.1016/j.ygyno.2015.09.078. Epub 2015 Sep 30. PMID 26428941
- [Background] Gallos ID, Shehmar M, Thangaratinam S, Papapostolou TK, Coomarasamy A, Gupta JK. Oral progestogens vs levonorgestrel-releasing intrauterine system for endometrial hyperplasia: a systematic review and metaanalysis. Am J Obstet Gynecol. 2010 Dec;203(6):547.e1-10. doi: 10.1016/j.ajog.2010.07.037. PMID 20934679
- [Derived] Alnemr AA, Harb OA, Atia H. The efficacy of the levonorgestrel intrauterine system versus oral megestrol acetate in treating atypical endometrial hyperplasia: a superior randomized controlled trial. J Gynecol Oncol. 2024 Sep;35(5):e62. doi: 10.3802/jgo.2024.35.e62. Epub 2024 Feb 22. PMID 38425141